CLINICAL TRIAL: NCT03810729
Title: Utility of a Smartphone Application in Assessing Palmar Circulation Prior to Radial Artery Harvesting for Coronary Artery Bypass Grafting
Brief Title: Smartphone Assessment Prior Radial Artery Harvesting for CABG
Acronym: iRADIAL-CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 20180865-01H
Record Dates: First submitted 2019-01-14; First posted 2019-01-22 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease
Keywords: Smartphone; Coronary artery bypass grafting; Modified Allen's Test
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Allen's Test (Active Comparator): The Modified Allen's Test (MAT) will be performed in a well-lit room on the participant's hand. This technique will involve compression of both the radial and ulnar arteries by the investigator to assess patency of the contralateral artery. The participant will then be asked to clench and open their hand several times. The participant will then be asked to maintain their hand in an open position. The investigator will then release the compression over the ulnar artery and observe for palmar blush. The length of time to achieve maximal palmar blush will be recorded. This technique will then be repeated by maintaining compression over the ulnar artery and releasing of the compression over the radial artery.
  Interventions: Diagnostic Test: Modified Allen's Test
- Smartphone assessment (Active Comparator): The smartphone app (Heart Rate, Azumio software) will be used to assess radial and ulnar artery patency. Briefly, the iPhone camera will be placed over the participant's index finger and patency assessed before and immediately following isolated contralateral artery compression for a maximum of two minutes.
  Interventions: Diagnostic Test: Smartphone assessment

INTERVENTIONS:
Diagnostic Test: Smartphone assessment — The smartphone app will be performed on participants randomly assigned to receive this test.
  Arms: Smartphone assessment
Diagnostic Test: Modified Allen's Test — The modified Allen's test will be will be performed on participants randomly assigned to receive this test.
  Arms: Modified Allen's Test

SUMMARY:
Coronary artery bypass graft (CABG) surgery is a procedure where surgeons use blood vessels from elsewhere in the body to go around blockages or narrowings in the heart arteries. Before the surgery, the surgeon needs to choose which vessel will be used for the bypass, including potentially the radial artery in the wrist. Smartphones have been shown in a previous study to be a better way to assess the arteries in the hand than the traditional physical examination, as it is less subjective than simply watching the flushing of the hand. In this study, the investigators will assess the utility of a smartphone application in determining whether there is enough blood flow in the hand prior to using the radial artery for CABG surgery.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is a procedure where surgeons use blood vessels from elsewhere in the body to go around blockages or narrowings in the heart arteries. Before the surgery, the surgeon needs to choose which vessel will be used for the bypass, including potentially the radial artery in the wrist. Before using this artery, it is important to ensure that there is enough blood flow to the hand to prevent complications. The best way to do this involves the use of ultrasound, but this takes a long time and its availability can be limited. Therefore, the assessment is usually done at the bedside by examining the hand, which relies on the doctor watching the flushing of the hand during compression and release of the artery. Currently, smartphones with cameras are able to assess blood flow by passing light through the skin and observing differences in brightness. This has been shown in a previous study to be a better way to assess the arteries in the hand than the traditional examination, as it is less subjective than simply watching the flushing of the hand. In this study, the investigators will assess the utility of a smartphone application in determining whether there is enough blood flow in the hand prior to using the radial artery for CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Scheduled to undergo coronary artery bypass graft for which the surgeon is considering the use of a radial artery conduit
* Able and willing to provide written informed consent

Exclusion Criteria:

* Hemodynamic instability
* Need for emergent cardiac surgery
* Known previous removal of the radial or ulnar arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with use of the radial artery as a conduit for CABG | In-hospital (average of 7 days)
  The primary outcome of this study is the use of the radial artery as a conduit in CABG surgery, which will only occur if the ulnar artery is deemed patent by the corresponding test to which the participant has been randomized to receive (i.e. modified Allen's test or smartphone assessment).

SECONDARY OUTCOMES:
Number of participants with post-operative hand ischemia | In-hospital (average of 7 days)
  Post-operative hand ischemia as determined by clinical assessment by attending physician or by need for a vascular intervention during index hospital admission.
Number of participants with early graft failure | In-hospital (average of 7 days)
  Early graft failure as determined by angiography during index hospitalization or by need for rescue percutaneous coronary intervention in the immediate post-operative period
Number of participants with stroke | In-hospital (average of 7 days)
  Stroke as determined by an attending neurologist
Number of participants with myocardial infarction | In-hospital (average of 7 days)
  Myocardial infarction as defined by the fourth universal definition of myocardial infarction.
Number of participants with cardiovascular death | In-hospital (average of 7 days)
  Death from cardiovascular cause as determined by attending physician.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hibbert, MD PhD, Principal Investigator — Ottawa Heart Institute Research Corporation; Vincent Chan, MD MPH, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data from the CAPITAL iRADIAL-CABG study will be made available upon a reasonable request to the principal investigator.
Time Frame: Data will be available following publication of our manuscript and will remain available for 10 years after this time.
Access Criteria: Access will be available upon a reasonable request to the principal investigator.

REFERENCES:
- [Derived] Goh CY, Parlow S, Di Santo P, Simard T, Jung R, Ahmed Z, Verreault-Julien L, Kuhar P, Chan V, Al-Atassi T, Toeg H, Bernick J, Wells GA, Ruel M, Hibbert B. Utility of a smartphone application in assessing palmar circulation prior to radial artery harvesting for coronary artery bypass grafting: rationale and design of the randomised CAPITAL iRADIAL-CABG trial. BMJ Open. 2022 Apr 8;12(4):e055580. doi: 10.1136/bmjopen-2021-055580. PMID 35396289